CLINICAL TRIAL: NCT03910478
Title: A Multi-Site, Randomized Trial of Subject-Collected Dried Blood Spot CMV Testing With Mobile Technology Support to Optimize Preemptive Therapy Late After Allogeneic HCT
Brief Title: Dried Blood Spot Testing of CMV Detection in HCT Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-0098; HHSN272201600015C
Record Dates: First submitted 2019-04-09; First posted 2019-04-10 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2021-01-04

CONDITIONS: Cytomegalovirus Infection
Keywords: Allogeneic; Cytomegalovirus; Dried Blood Spot; Hematopoietic cell transplantation
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Self-collected Dried Blood Spot (DBS) monitoring (Experimental): N=100 Subject collected DBS CMV monitoring with mobile technology support
  Interventions: Device: DBS Self-Collection Kit
- Standard Monitoring Control (Active Comparator): N=50 Standard care with office based testing
  Interventions: Other: Standard Control Strategy

INTERVENTIONS:
Device: DBS Self-Collection Kit — Kit for self-collection of Dried Blood Spot (DBS) samples
  Arms: Self-collected Dried Blood Spot (DBS) monitoring
Other: Standard Control Strategy — Standard of care with office-based testing.
  Arms: Standard Monitoring Control

SUMMARY:
This is a randomized clinical trial to assess whether a subject centered, self-collection of Dried blood spots (DBS) samples will improve compliance with the clinical recommendation of weekly Cytomegalovirus (CMV) testing of Hematopoietic cell transplantation (HCT) recipients who are at high risk for late CMV disease. In this study, mobile devices will be used to remind HCT survivors to perform CMV monitoring using finger-stick collected DBS testing in their home setting or to visit their doctor's office to perform the test. 150 allogeneic HCT recipients > /= 15 years of age will be randomized (2:1) to DBS monitoring or standard of care (per local institution) monitoring. Duration of study participation is anticipated to be within a range of 26 weeks to 43 weeks. The primary objective is to evaluate adherence to recommended CMV monitoring duration and interval during the first year after HCT upon enrollment using subject collected dried blood spot testing.

DETAILED DESCRIPTION:
This is a randomized clinical trial to assess whether a subject centered, self-collection of dried blood spots (DBS) samples will improve compliance with the clinical recommendation of weekly Cytomegalovirus (CMV) testing of Hematopoietic cell transplantation (HCT) recipients who are at high risk for late CMV disease. In this study, mobile devices will be used to remind HCT survivors to perform CMV monitoring using finger-stick collected DBS testing in their home setting or to visit their doctor's office to perform the test. 150 allogeneic HCT recipients > /= 15 years of age will be randomized (2:1) to DBS monitoring or standard of care (per local institution) monitoring. Duration of study participation is anticipated to be within a range of 26 weeks to 43 weeks. The primary objective is to evaluate adherence to recommended CMV monitoring duration and interval during the first year after HCT upon enrollment using subject collected dried blood spot testing. The secondary objectives are 1) To evaluate the mean difference between the recommended monitoring that each subject completes between the DBS and the control arm. 2) To compare the incidence of CMV disease between the DBS monitoring and standard of care arm; 3) To evaluate the safety of DBS monitoring.

Additionally, an observational cohort of 450 HCT recipients, who consented for retrospective studies and meet eligibility criteria but are not participating in the DBS testing for CMV, will be used to assess whether randomized study sample is representative of the DBS study population and to obtain a population-based estimate of late CMV disease.

ELIGIBILITY:
Inclusion Criteria:

Randomized Cohort:

1. Must be >/= 15 years of age at the time of enrollment
2. Must be able to provide written consent and complete the informed consent
3. Must have received allogeneic hematopoietic cell transplantation within 60-180 days prior to randomization
4. Cytomegalovirus (CMV) seropositive or had a donor who was CMV positive
5. One or both of the following:

   * CMV event* within the first 100 days post-transplant requiring anti-viral treatment
   * Receipt of CMV prophylaxis**(for at least 30 days) prior to randomization. Continuation of letermovir or acyclovir/valacyclovir (high and low dose) prophylaxis after day 100 per institutional standard of care is permitted * CMV event defined as deoxyribonucleic acid (DNA) detection or disease ** Anti-viral treatment or prophylaxis includes ganciclovir, valganciclovir, foscarnet, letermovir, maribavir or acyclovir/valacyclovir (high and low dose)
6. Direct availability to the internet either by a computer in the residence or a smart phone
7. Had at least one or more of these conditions:

   * HLA mismatch*
   * umbilical cord blood source**
   * Graft versus host disease (GVHD)***
   * T-cell depletion**** * Human leukocyte antigen (HLA)-related (sibling) donor with at least one mismatch at one of the following three HLA-gene loci: HLA-A, -B, or -DR, Haploidentical donor, Unrelated donor with at least one mismatch at one of the following four HLA-gene loci: HLA-A, -B, -C and -DRB1

     * Use of umbilical cord blood as stem cell source ***Acute or chronic GVHD requiring topical steroid for gastrointestinal (GI) GVHD and/or systemic steroid treatment (>/= 1 mg/kg/day of prednisone or equivalent dose of another corticosteroid) within 6 weeks prior to enrollment

       * Subjects who have received partial or full T-cell depletion (with or without GVHD). T-cell depletion can be given as either ex-vivo or in-vivo for GVHD prophylaxis. T-cell depleting agents include, but are not limited to, anti-thymocyte globulin (ATG) and alemtuzumab

Observation Cohort:

1. Must be >/= 15 years of age at the time of enrollment
2. Must have one of the following:

   * Consented for retrospective studies at their transplant center, or
   * Be included under the auspices of the site's IRB approved waiver of additional consent for retrospective studies
3. Must have received allogeneic hematopoietic cell transplantation during or within 1 year prior to the conduct of the randomized trial (defined as time during which randomization is done)
4. CMV seropositive or had a donor who was CMV positive
5. One or both of the following:

   * CMV event* within the first 100 days post-transplant requiring anti-viral treatment
   * Receipt of CMV prophylaxis**(for at least 30 days) prior to registration. Continuation of letermovir prophylaxis or acyclovir/valacyclovir (high and low dose) after day 100 per institutional standard of care is permitted * CMV event defined as DNA detection or disease ** Anti-viral treatment or prophylaxis includes ganciclovir, valganciclovir, foscarnet, letermovir, maribavir or acyclovir/valacyclovir (high and low dose)
6. Meet at least one or more of criteria of the following:

   * HLA mismatch*
   * umbilical cord blood source**
   * GVHD***
   * T-cell depletion****

     * Human leukocyte antigen (HLA)-related (sibling) donor with at least one mismatch at one of the following three HLA-gene loci: HLA-A, -B, or -DR, Haploidentical donor, Unrelated donor with at least one mismatch at one of the following four HLA-gene loci: HLA-A, -B, -C and -DRB1

       * Use of umbilical cord blood as stem cell source ***Acute or chronic GVHD requiring topical steroid for GI GVHD and/or systemic steroid treatment (>/= 1 mg/kg/day of prednisone or equivalent dose of another corticosteroid) within 6 weeks prior to enrollment ****Subjects who have received partial or full T-cell depletion (with or without GVHD). T-cell depletion can be given as either ex-vivo or in-vivo for GVHD prophylaxis. T-cell depleting agents include, but are not limited to, anti-thymocyte globulin (ATG) and alemtuzumab

Exclusion Criteria:

Randomized Cohort:

1. Inability to fully comprehend the study website and study procedures
2. Any other condition, which in the opinion of the investigator would interfere with successful completion of this clinical trial
3. Morphological relapse (bone marrow or peripheral blood blast) prior to registration

Observational Cohort:

1. Did not meet all inclusion criteria
2. Morphological relapse (bone marrow or peripheral blood blast) prior to registration

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Minnesota Medical Center, Fairview - Infectious Diseases and International Medicine, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The University of Texas - MD Anderson Cancer Center - Infectious Diseases, Houston, Texas
  - Fred Hutchinson Cancer Research Center - Vaccine and Infectious Diseases, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were considered by their transplant teams to be at risk for late CMV disease and were clinically recommended to continue CMV monitoring after day 100 post-transplant were recruited from 4 clinical sites within the United States. The first participant was enrolled on May 3, 2019 and the last participant was enrolled on July 27, 2023.
Groups:
- Self-collected Dried Blood Spot (DBS) Monitoring: Participants collected DBS CMV monitoring with mobile technology support.
  DBS Self-Collection Kit: Kit for self-collection of Dried Blood Spot (DBS) samples.
- Standard Monitoring Control: Standard care with office based testing.
  Standard Control Strategy: Standard of care with office-based testing.
Period: Overall Study
Arm/Group | Self-collected Dried Blood Spot (DBS) Monitoring | Standard Monitoring Control
Started | 113 | 59
Completed | 68 | 51
Not Completed | 45 | 8
Not completed — Death | 13 | 6
Not completed — Withdrawal by Subject | 23 | 2
Not completed — Physician Decision | 5 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Failure to meet continuation criteria | 2 | 0
Not completed — Wouldn't proceed DBS portion, data collection only | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-collected Dried Blood Spot (DBS) Monitoring | Standard Monitoring Control | Total
Number analyzed (Participants) | 113 | 59 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (14.4) | 49.7 (16.0) | 52.2 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 30 | 69
  Male | 74 | 29 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 20
  Not Hispanic or Latino | 100 | 48 | 148
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 10 | 4 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 4 | 14
  White | 83 | 42 | 125
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 6 | 6 | 12
Transplant Site [Count of Participants; unit: Participants]
  Fred Hutchinson Cancer Research Center | 34 | 18 | 52
  Memorial Sloan Kettering Cancer Center | 19 | 8 | 27
  University of Minnesota Medical School | 22 | 13 | 35
  MD Anderson Cancer Center | 38 | 20 | 58
Perceived Ease of Access to Blood Draw Facility [Count of Participants; unit: Participants]
  Easy | 97 | 51 | 148
  Difficult | 16 | 8 | 24
Days from HCT [Mean (Standard Deviation); unit: days] | 88.6 (24.4) | 86.2 (15.4) | 87.8 (21.7)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Have Completed >90% of Their Recommended Cytomegalovirus (CMV) Monitoring Tests in the DBS and Control Arms in the ITT Population
Description: To evaluate adherence to recommended CMV monitoring duration and interval during the first year after HCT, the number of participants who completed >90% of their recommended CMV monitoring tests at one year after HCT in the DBS and control arms was collected.
Time Frame: At one year after Hematopoietic cell transplantation (HCT)
Population: The Intention-to-Treat population (ITT) included all participants in the randomized cohort in the intervention group to which they were randomly assigned, regardless of their monitoring compliance and regardless of subsequent withdrawal or deviation from the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-collected Dried Blood Spot (DBS) Monitoring | Standard Monitoring Control
Number analyzed (Participants) | 113 | 59
Participants | 27 | 15
Statistical Analysis 1: Comparison: Self-collected Dried Blood Spot (DBS) Monitoring vs Standard Monitoring Control; A traditional logistic regression model was fit where the outcome was whether or not participants completed > 90% of their clinician-recommended CMV monitoring tests in the study period by 1-year after HCT; Test type: Equivalence — A two-sided Wald-test for evidence of a non-zero coefficient for intervention group in the regression was conducted at the 5% significance level; p = 0.8920, Regression, Logistic; The logistic regression was adjusted by covariates (transplant site and participant's perceived ease of access to blood draw facility); Odds Ratio (OR) = 0.948, 95% CI 2-sided [0.438 to 2.053]

2. Primary Outcome: The Number of Participants Who Have Completed >90% of Their Recommended Cytomegalovirus (CMV) Monitoring Tests in the DBS and Control Arms in the mITT Population
Description: as for outcome 1
Time Frame: At one year after Hematopoietic cell transplantation (HCT)
Population: The mITT population included all participants in the ITT population who had at least one result for the number of clinician-recommended CMV monitoring tests and remained enrolled through their first scheduled clinician recommended CMV monitoring test. Participants were grouped based on the intervention received, where participants that completed at least one self-collected DBS sample were grouped in the DBS arm and all other participants were grouped in the SOC arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-collected Dried Blood Spot (DBS) Monitoring | Standard Monitoring Control
Number analyzed (Participants) | 82 | 63
Participants | 22 | 20
Statistical Analysis 1: Comparison: Self-collected Dried Blood Spot (DBS) Monitoring vs Standard Monitoring Control; A traditional logistic regression model was fit where the outcome was whether or not participants completed > 90% of their clinician -recommended CMV monitoring tests in the study period by 1-year after HCT; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.3008, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.660, 95% CI 2-sided [0.301 to 1.450]

3. Secondary Outcome: The Total Number of Recommended Cytomegalovirus (CMV) Monitoring Tests That Were Completed Per Participant in the ITT Population
Description: The total number of recommended Cytomegalovirus (CMV) monitoring tests that were completed per participant was reported.
Time Frame: By 1 year after Hematopoietic cell transplantation (HCT)
Population: as for outcome 1
Measure: Median (Full Range); unit: number of monitoring tests completed
Arm/Group | Self-collected Dried Blood Spot (DBS) Monitoring | Standard Monitoring Control
Number analyzed (Participants) | 113 | 59
number of monitoring tests completed | 6 [0 to 45] | 11 [0 to 55]

4. Secondary Outcome: The Total Number of Recommended Cytomegalovirus (CMV) Monitoring Tests That Were Completed Per Participant in the mITT Population
Description: The total number of recommended Cytomegalovirus (CMV) monitoring tests that were completed per participant was reported.
Time Frame: By 1 year after Hematopoietic cell transplantation (HCT)
Population: as for outcome 2
Measure: Median (Full Range); unit: number of monitoring tests completed
Arm/Group | Self-collected Dried Blood Spot (DBS) Monitoring | Standard Monitoring Control
Number analyzed (Participants) | 82 | 63
number of monitoring tests completed | 11 [0 to 45] | 11 [0 to 55]

5. Secondary Outcome: Number of Participants With End-organ Cytomegalovirus (CMV) Disease, Possible and Proven/Probable
Description: Proven or probable CMV disease is a serious adverse event of special interest. The number of participants experiencing proven or probable CMV disease between Hematopoietic cell transplantation (HCT) and 365 days after HCT.
Time Frame: By 1 year after Hematopoietic cell transplantation (HCT)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Self-collected Dried Blood Spot (DBS) Monitoring | Standard Monitoring Control
Number analyzed (Participants) | 113 | 59
Participants
  Possible | 0 | 0
  Probable | 0 | 0
  Proven | 2 | 2
  Probable/Proven | 2 | 2

6. Secondary Outcome: Number of Participants With Finger-stick Procedure-related Grade 3 Adverse Events (AEs) in the DBS Arm
Description: To evaluate the safety of DBS monitoring, Finger-stick procedure-related Grade 3 AEs were abstracted through medical chart review at quarterly contacts and at the final close-out contact. Participants were considered as meeting the outcome measure if they had at least one finger-stick procedure-related Grade 3 AE during the study period.
Time Frame: By 1 year after Hematopoietic cell transplantation (HCT)
Population: The safety population consist of all enrolled participants that had any safety data collected after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-collected Dried Blood Spot (DBS) Monitoring
Number analyzed (Participants) | 94
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of Hematopoietic cell transplantation (HCT) to 365 days after HCT (final study visit).
Description: All-Cause Mortality was collected for all randomized participants. AEs were assessed differently depending on analysis population and study arm. SAEs of special interest (proven/probable CMV disease) were collected for all participants in the Safety Population. Other AEs considered severe and related to the DBS collection and finger stick procedure were collected for participants in the Safety Population in the DBS arm only; no other AEs were collected in the Standard Monitoring Control Arm.
Arm/Group | Self-collected Dried Blood Spot (DBS) Monitoring | Standard Monitoring Control
All-Cause Mortality (participants affected / at risk) | 16/113 | 7/59
Serious Adverse Events (participants affected / at risk) | 2/94 | 2/58
Other Adverse Events (participants affected / at risk) | 0/94 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self-collected Dried Blood Spot (DBS) Monitoring (N=94) | Standard Monitoring Control (N=58)
Cytomegalovirus gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus duodenitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT03910478/Prot_001.pdf
  • Statistical Analysis Plan (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT03910478/SAP_002.pdf
  • Informed Consent Form (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT03910478/ICF_000.pdf